# Statistical Analysis Plan

**Protocol No. MT-1186-Z-101** 

A Phase I, Randomized, Open-Label, Crossover-Design, Single-Dose Study to Investigate the Safety, Tolerability and Comparative Bioavailability of Oral Edaravone Administered orally and via a Nasogastric Tube (NGT) in Healthy Adult Subjects

| Prepared By: | |
|--------------|-----------|
| Version: | Ver1.0 |
| Date: | 22JUN2021 |

NCT number: NCT04776135

#### APPROVAL FORM

Statistical Analysis Plan

| Protocol No. | MT-1186-Z-101 |
|---|---|
| Protocol Title | A Phase I, Randomized, Open-Label, Crossover-Design, Single-Dose Study to Investigate the Safety, Tolerability and Comparative Bioavailability of Oral Edaravone Administered orally and via a Nasogastric Tube (NGT) in Healthy Adult Subjects |
| Version / Date | V1.0 / 22JUN2021 |

#### **Authors:**

| Statistics / Clinical Pha | rmacokinetics A | uthor |
|---------------------------|-----------------|-------|
| Print Name: | | |
| Position: | | |

# Reviewed by:

| Statistic reviewer | of MTPC |
|--------------------|---------------------------|
| Print Name: | |
| Position: | COT STAT |
| Clinical Pharmaco | okinetic reviewer of MTPC |
| Print Name: | |
| Position: | СОТ СР |

# Approved by:

| Statistic / Clinical Phan | macokinetic A ver |
|---------------------------|-----------------------|
| Print Name: | |
| Position: | Head of STA |
| Signature: | |
| Approval date: | |
| Statistic Approver of M | TPC |
| Print Name: | |
| Position: | Responsible STAT |
| Signature: | |
| Approval date: | |
| Clinical Pharmacokine | tic Approver of MTPC_ |
| Print Name: | |
| Position: | Responsible CP |
| Signature: | |
| Approval date: | |

Confidential

# TABLE OF CONTENTS

| Introduction | |
|--------------------------------------------------------|-----|
| 2 Study Objective and Endpoints | . 8 |
| 2.1 Study Objective(s) | . 8 |
| 2.1.1 Safety Assessment(s) | . 8 |
| 2.1.2 Pharmacokinetics Assessment(s) | . 8 |
| 3 Study Design | . 9 |
| 3.1 Phase and Type of the Study | . 9 |
| 3.2 Study Design | . 9 |
| 3.2.1 Type and Details of Cohorts | . 9 |
| 3.2.2 Study Period and Evaluation Period | . 9 |
| 3.3 Schedule of Study Procedures | |
| 3.4 Sample Size and Power Considerations | |
| 4 Planned analysis | |
| 4.1 Final Analysis | |
| 5 Analysis populations | |
| 6 Statistical considerations | |
| 6.1 Descriptive Statistics | 15 |
| 6.2 Statistical Tests and Estimates | .15 |
| 7 Data Conventions | |
| 7.1 Analysis Variable Definitions | |
| 7.1.1 Study Subjects | |
| 7.1.1.1 Demographic and Other Baseline Characteristics | .16 |
| 7.1.1.2 Medical History | |
| 7.1.1.3 Concomitant Medication | |
| 7.1.2 Safety Assessments | |
| 7.1.2.1 Adverse Events | |
| 7.1.2.2 Laboratory Tests | |
| 7.1.2.3 12-Lead ECG | |
| 7.1.3 Pharmacokinetics Evaluation | |
| 7.1.3.1 Plasma Concentration | |
| 7.1.3.2 Pharmacokinetic Parameters | |
| | .19 |
| 7.3 Data Handling Convention for Missing Data | .20 |
| 8 Statistical Methodology | |
| 8.1 Study Subjects | |
| 8.1.1 Subject Disposition | |
| 8.1.2 Analysis Populations | |
| 8.1.3 Study Drug Exposure | |
| 8.1.4 Demographic and Other Baseline Characteristics | .21 |
| 8.1.5 Medical History | .22 |
| 8.1.6 Concomitant Medications | |
| 8.2 Safety Assessments | |
| 8.2.1 Adverse Events | |
| 8.2.2 Laboratory Tests | |
| 8.2.3 Vital Signs | .23 |
| 0.2.0 | |

| Statistical Analysis Plan Protocol No. MT-1186-Z-101 | Aitsubishi Tanabe Pharma Corporation |
|---|---|
| 8.2.4 12-Lead ECGs | 24 |
| 8.2.5 Physical Examinations | |
| 8.3 Pharmacokinetics Evaluation | |
| 8.3.1 Plasma Concentrations and Pharmacokinetic Parame | eters24 |
| 8.3.2 Pharmacokinetic Parameters | |
| 8.3.3 Analysis of Variance | |
| 9 Data Presentation Conventions | |
| 9.1 Number of Digits to Report | 26 |
| 9.2 Treatments and Groups to Report | 27 |
| 9.3 Period, Visit and Time Point to Report | |
| 10 Change from the Protocol | |
| 11 Software | 30 |
| 12 References | |
| Appendix 1 Pharmacokinetic Parameter Calculations | |

# **ABBREVIATIONS**

| Abbreviations | Definitions |
|---------------|----------------------------------------------|
| AE | adverse event |
| ALS | amyotrophic lateral sclerosis |
| ALT | alanine transaminase |
| ALP | alkaline phosphatase |
| ANOVA | analysis of variance |
| APTT | activated partial thromboplastin time |
| AST | aspartate transaminase |
| BLQ | below limit of quantification |
| BMI | body mass index |
| CI | confidence interval |
| CK | creatine phosphokinase |
| CRP | c-reactive protein |
| CV | coefficient of variation |
| DP | decimal places |
| ECG | electrocardiogram |
| γ-GTP | γ-glutamyltranspeptidase |
| HDL | High-density lipoprotein |
| INR | prothrombin international normalized ratio |
| LDH | lactate dehydrogenase |
| LDL | low-density lipoprotein |
| LLOQ | lower limit of quantitation |
| LOQ | limit of quantification |
| LS | least square(s) |
| MedDRA | medical dictionary for regulatory activities |
| MTPC | Mitsubishi Tanabe Pharma Corporation |
| NGT | Nasogastric Tube |
| PK | pharmacokinetics |
| PKPOP | PK Population |
| PO | per os |
| PT | preferred term |
| QTcF | fridericia's correction of QT interval |
| RBC | red blood cell |
| SAP | statistical analysis plan |
| SAE | serious adverse event |
| SAF | safety population |
| SD | standard deviation |
| SOC | system organ class |
| WBC | white blood cell |
| WHO | World Health Organization |

# LIST OF PK PARAMETERS

| Parameters | Unit | Definitions |
|---|---|---|
| AUC <sub>0-24</sub> | ng•h/mL | Area under the plasma concentration-time curve from zero up to 24 hours |
| AUC <sub>0-t</sub> | ng•h/mL | Area under the plasma concentration-time curve from zero up to the last quantifiable concentration time point |
| AUC <sub>0-∞</sub> | ng•h/mL | Area under the plasma concentration-time curve from zero up to infinity with extrapolation of the terminal phase |
| AUC% <sub>ex</sub> | % | Area under the (plasma) concentration-time curve extrapolated from the last quantifiable concentration time point to infinity in % of the total AUC <sub>0-∞</sub> |
| $C_{max}$ | ng/mL | Maximum plasma concentration after administration |
| CL/F | L/h | Apparent total clearance |
| $k_{\rm el}$ | 1/h | Elimination rate constant from the central compartment |
| MRT | h | Mean residence time |
| t <sub>1/2</sub> | h | Terminal elimination half-life in plasma concentration-time course |
| $t_{ m max}$ | h | Time of C <sub>max</sub> |
| V <sub>ss</sub> /F | L | Apparent volume of distribution at steady state |
| V <sub>z</sub> /F | L | Apparent volume of distribution during terminal phase |

#### 1 INTRODUCTION

This statistical analysis plan (SAP) is based on the final protocol (01.01.00000) dated 12-Feb-2021. The plan covers statistical analysis, tabulations and listings of the study data to investigate the pharmacokinetics and safety.

Any statistical analysis details described in this document supersede any description of statistical analysis in the protocol.

#### 2 STUDY OBJECTIVE AND ENDPOINTS

#### 2.1 Study Objective(s)

Primary objective:

To investigate the comparative bioavailability of edaravone oral suspension administered orally and via a nasogastric tube in healthy adult subjects

Secondary objective:

To investigate the pharmacokinetics, safety, and tolerability of a single dose of edaravone oral suspension in healthy adult subjects

#### 2.1.1 Safety Assessment(s)

- (1) Adverse events (AEs) and adverse drug reactions (ADRs)
- (2) 12-lead ECG
- (3) Laboratory tests
- (4) Vital signs

#### 2.1.2 Pharmacokinetics Assessment(s)

(1) Drug concentration (in plasma)

Unchanged edaravone

(2) Pharmacokinetic parameters

AUC<sub>0-t</sub> (t: Final time point when concentration is measurable), AUC<sub>0-∞</sub>,  $C_{max}$ , AUC<sub>0-24</sub>,  $t_{max}$ ,  $t_{1/2}$ ,  $k_{el}$ , MRT, CL/F,  $V_z/F$ , and  $V_{ss}/F$ .

#### 3 STUDY DESIGN

#### 3.1 Phase and Type of the Study

Phase of the study

: Phase I

Type of the study

: Clinical pharmacology study

#### 3.2 Study Design

#### 3.2.1 Type and Details of Cohorts

Single-dose, randomization, open-label, crossover study.

| Group (number of subjects) | Period I | Period II |
|---|---|---|
| Oral administration precedent | Oral administration of edaravone oral suspension | Nasogastric administration of edaravone oral suspension |
| (18 subjects) | 105 mg | 105 mg |
| NItwin odministration | Nasogastric administration of | Oral administration of |
| Nasogastric administration precedent (18 subjects) | edaravone oral suspension | edaravone oral suspension |
| precedent (18 subjects) | 105 mg | 105 mg |

Thirty-six subjects are randomly allocated to two groups of 18 subjects. It is carried out by the two-period, two-sequence crossover, randomization, open-label study. The duration of hospitalization will be 7 days and 6 nights.



#### 3.2.2 Study Period and Evaluation Period

Study period: The study period is defined as the period from the time of obtaining the informed consent to the time of completion of the end-of-study assessment or discontinuation assessment (for subjects who entered the follow-up period, to the time of completion or termination of the follow-up).

Statistical Analysis Plan Protocol No. MT-1186-Z-101

Mitsubishi Tanabe Pharma Corporation

Screening: Subjects providing informed consent were screened for eligibility to select subjects meeting all of the inclusion criteria and none of the exclusion criteria (36 subjects with a few reserve subjects).

Evaluation period: The evaluation period is defined as the period from completion of dosing of the investigational product in Period I to completion of the end-of-study assessment or discontinuation assessment.

End-of-study assessment: The prespecified observations and tests were performed as the end-of-study assessment, 7 days (±2 days) after the last dose of the investigational product.

Mitsubishi Tanabe Pharma Corporation

# 3.3 Schedule of Study Procedures

| | Informed | Screening | | | | | | | п. | Period I | 90 | _ | | ı | ı | | | | | | | | | | | 111 | Peri | Period I | _ | | | | | | | End-of-study <sup>a)</sup><br>Assesment | in dy |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day (time window) | consent | Day -30<br>to -2 | 7 | | | | | | <b>-</b> | _ | | | | | | | ~ | 2 | 3 | | | | | | | 4 | | | } | | - | } | | ro. | 9 | 11 (±2) | |
| Time after dosing | | Visit | Pre-dose<br>Admission | O Dra doco | 5 m | 15 m | 30 m | 45 m | 1 h | 1 h 30 m | 2 h | 4 h | 6 h | 8 h | 10 h | 12 h | 24 h | 36 h | 48 h | Pre-dose | 0 | 5 m | 15 m | 30 m | 45 m | 1 h | 1 h 30 m | 2 h | 4 h | 6 h | 10 h<br>8 h | 12 h | 24 h | 36 h | 48 h | Visit | |
| Screening | | × | $\vdash$ | $\vdash$ | Н | Ш | Ц | | | | | | | | | | | | | | | | | | $\dashv$ | | $\dashv$ | 7 | $\dashv$ | - | _ | - | - | 4 | 4 | | |
| Written informed consent | × | | Н | | | | | | | | | | | | | | | | $\Box$ | | | | | $\dashv$ | $\dashv$ | $\dashv$ | $\dashv$ | $\dashv$ | $\dashv$ | $\dashv$ | $\dashv$ | $\dashv$ | $\dashv$ | | - | | |
| Subject characteristics | | × | Н | | $\vdash$ | | Ц | | | | | | | | | | | $\Box$ | | | | | | _ | 7 | $\dashv$ | 7 | $\dashv$ | $\dashv$ | + | - | $\dashv$ | $\dashv$ | 4 | 4 | | |
| Eligibility assessment | | × | × | ال | - | $\sqcup$ | _ | | | | | | | | | ╗ | | | | | | | | 7 | + | 7 | $\dashv$ | 7 | + | $\dashv$ | $\dashv$ | $\dashv$ | $\dashv$ | + | 4 | | |
| Nasal Examination | | × | | | $\dashv$ | | Ц | | | | | | | | | | | | | | | | | $\exists$ | 1 | 寸 | | $\dashv$ | $\dashv$ | $\dashv$ | $\dashv$ | $\dashv$ | $\dashv$ | + | $\dashv$ | | |
| Height | | × | | | | | | | | | | | | | | | | | | | | | | $\dashv$ | $\dashv$ | $\dashv$ | $\dashv$ | + | - | $\dashv$ | $\dashv$ | $\dashv$ | $\dashv$ | + | | | |
| Weight | | × | × | H | Н | | | | | | | | | | | | | | | | | | | $\dashv$ | $\dashv$ | 寸 | 寸 | $\dashv$ | $\dashv$ | + | $\dashv$ | $\dashv$ | $\dashv$ | $\dashv$ | $\dashv$ | × | |
| BMI | | × | × | H | | | | | | | | | | | | | | | | | | | | 7 | 7 | 寸 | $\dashv$ | $\dashv$ | - | 7 | $\dashv$ | $\dashv$ | $\dashv$ | + | 4 | | |
| Physical examination | | × | X | - | | | | | × | | | | | | | | × | | × | × | | | | | | × | • | | | _ | $\dashv$ | - | <del>^</del> | × | × | | |
| Vítal signs | | × | × | <u>_</u> | $\vdash$ | _ | | | Х | | | | | | | | × | | × | × | | | | | | × | $\dashv$ | $\dashv$ | $\dashv$ | $\dashv$ | $\dashv$ | $\dashv$ | ∸∣ | 닔 | ×۱ | × | |
| 12-lead ECG | | × | × | ٦ | $\vdash$ | _ | | | X | | | | | | | | × | | × | × | | | | | $\dashv$ | × | $\dashv$ | $\dashv$ | $\dashv$ | $\dashv$ | $\dashv$ | ┥ | × | ᅴ | × | | |
| Laboratory tests | | × | × | Н | Н | Н | | | | | | | | | | | | | × | | | | J | ╗ | $\neg$ | | $\dashv$ | $\dashv$ | $\dashv$ | | | $\dashv$ | + | + | × | × | |
| Serological tests | | × | | $\dashv$ | $\dashv$ | | _ | | | | | | | | | | | | | $\Box$ | | | | | 7 | $\dashv$ | 7 | $\dashv$ | + | + | $\dashv$ | $\dashv$ | $\dashv$ | $\dashv$ | _ | | |
| Drug/alcohol abuse screening | | × | | | | | | | | | | | | | | | | | | | | | | ╗ | ┪ | ╛ | 一 | $\dashv$ | -1 | ᅥ | $\dashv$ | $\dashv$ | ᅥ | $\dashv$ | | | |
| Pregnancy test in female | | × | × | $\vdash$ | $\vdash$ | $\sqcup$ | Ц | | | | | | | | | | | | $\Box$ | $\Box$ | | | | | 1 | $\exists$ | $\exists$ | 1 | $\dashv$ | $\dashv$ | + | - | + | $\dashv$ | _ | × | |
| COVID-19 virus test | | | × | | | | | | | | | | | | | | | | | | | | | | $\dashv$ | $\dashv$ | $\exists$ | | - | $\dashv$ | $\dashv$ | - | $\dashv$ | $\dashv$ | - | | |
| Dosing of edaravone | | | Н | $\exists$ | × | $\sqcup$ | Ц | | | | | | | | | | | | | | × | | | | ┪ | ╛ | ┪ | ┪ | $\dashv$ | 1 | $\dashv$ | - | $\dashv$ | $\dashv$ | - | | |
| Adverse events <sup>b)</sup> | V | | + | + | + | + | + | | $\int$ | | | Ľ | Ī | | $oldsymbol{\mathbb{L}}$ | Ι | | | Ц | Ц | | $\prod$ | | Ħ | $\dagger \dagger$ | $\dagger \dagger$ | $\dagger \dagger$ | $\dagger \dagger$ | $\dagger \dagger$ | $\parallel$ | H | Н | ╫ | H | $\mathbb{H}$ | | $\uparrow$ |
| Concomitant medications | | | $\downarrow$ | + | + | $\mathbb{H}$ | Щ | Ш | | | | $\perp$ | Ц | П | Ш | | $\prod$ | Ш | Ш | Щ | | $\prod$ | | Ħ | П | П | $\dagger \dagger$ | $\dagger \dagger$ | $\dagger$ | $\forall$ | H | ╫ | Н | H | $\mathbb{H}$ | | $\uparrow$ |
| PK Blood sampling for edaravone | | | × | 닛 | × | × | × | × | × | × | × | $\ge$ | × | × | × | × | × | × | × | × | ╝ | × | × | × | × | × | × | × | × | × | × | $\stackrel{\sim}{\sim}$ | $\stackrel{\sim}{\sim}$ | × | 끩 | | |

<sup>4)</sup> At the time of withdrawal, perform the same tests as would be performed in the end-of-study assessment.

(b) Collecting serious adverse events was started after informed consent was obtained. Collecting the other adverse events was started after informed consent was obtained. Collecting the other adverse events was started after informed consent was obtained.

#### 3.4 Sample Size and Power Considerations

Total of 36 subjects

#### [Rationales for setting]

A sample size of 36 subjects was set to ensure 30 completing subjects allowing for 6 dropouts based on the results of a bioavailability study of TIGLUTIC® (Riluzole suspension) administered orally versus NGT administration (Benjamin Rix Brooks et al., 2019) and practical experiences in preceding studies.

#### 4 PLANNED ANALYSIS

#### 4.1 Final Analysis

This SAP will be finalized before database lock. Final data analysis will be performed after database lock.

#### 5 ANALYSIS POPULATIONS

Pharmacokinetic (PK) analysis will be performed on the PK analysis set (PKPOP). Safety analysis will be performed on the safety analysis set (SAF). The definitions of the analysis sets are provided below. The detailed handling of subjects will be determined by the sponsor, by the time of database lock.

#### (1) PK analysis set (PKPOP)

The PK analysis set will consist of all subjects who received at least 1 dose of the investigational product and have evaluable PK data.

## (2) Safety analysis set (SAF)

The SAF will consist of all subjects who received at least 1 dose of the investigational product.

#### 6 STATISTICAL CONSIDERATIONS

#### 6.1 Descriptive Statistics

#### (1) Non-PK related

Continuous data will be summarized descriptively using the number in the analysis set (N), the number of observations (n), mean, SD, median, minimum and maximum. Categorical data will be summarized using frequency counts and percentages. The denominator for the percentages will be the total number of subjects in the treatment/group and analysis population applied, unless otherwise specified.

#### (2) PK related

#### 1) Plasma concentrations

Plasma concentrations will be summarized descriptively using N, n, mean, SD, CV%, median, minimum and maximum.

#### 2) Pharmacokinetic parameters

The plasma PK parameters will be summarized descriptively using N, n, mean (i.e. arithmetic mean), SD, CV%, median, minimum, maximum, geometric mean and geometric CV%.

CV% and Geometric CV% will be calculated as follows:

$$CV\% = \frac{SD}{arithmetic mean} \times 100$$

Geometric CV% = 
$$\sqrt{[\exp(\sigma^2) - 1]} \times 100$$

where  $\sigma$  represents the SD calculated from the natural logarithmic transformed value of parameters.

#### 6.2 Statistical Tests and Estimates

No statistical tests will be performed. Confidence level will be 0.90, so that two-sided 90% CIs will be calculated where applicable.

#### 7 DATA CONVENTIONS

# (1) Handling of data for PK assessments

If it is necessary to investigate the data handling because of, for example, a protocol deviation (e.g., the blood collection time fell outside the allowable range, the plasma drug concentration could not be measured, or the blood plasma collection procedures were not followed), the study sponsor will decide on the data handling. PK data that are considered "invalid" will be flagged as such in the data listings and will not be included in the summary tables and figures. These data can be excluded from calculation of PK parameters. The PK data handling will be assessed at the data review meeting prior to database lock and a document for PK data handling will be issued.

#### 7.1 Analysis Variable Definitions

#### 7.1.1 Study Subjects

#### 7.1.1.1 Demographic and Other Baseline Characteristics

(1) BMI

BMI will be recalculated using the formula below and reported to 1 DP.

BMI  $(kg/m^2)$  = weight at Day -1 (kg) / {height at screening (m)}<sup>2</sup>

#### 7.1.1.2 Medical History

Medical history will be coded according to the MedDRA version 23.1. Definitions of categories are as follows:

#### (1) Medical history

Any medical conditions which had stopped before the first administration of investigational product.

#### (2) Complication

Any medical conditions which were present at the first administration of investigational product.

#### (3) Allergic history

Medical conditions which were reported as allergic history.

#### 7.1.1.3 Concomitant Medication

Medications will be coded according to the WHO (WHO) Drug Global B3 Format September 1, 2020.

Concomitant medication is any medication (including commercially available drugs) other than the investigational product, used between the first administration of investigational product and completion of the end-of-study assessment.

#### 7.1.2 Safety Assessments

#### 7.1.2.1 Adverse Events

Adverse events will be coded according to the MedDRA version 23.1.

#### (1) Adverse Events (AEs)

An AE is any untoward medical occurrence or unintended sign (including an abnormal laboratory finding), symptoms and disease, occurred after administration and observed in the safety assessment period, regardless of causal relationship with the investigational product. However, if an existing AE worsens in grade or severity, it will be treated as a new AE.

#### (2) Serious Adverse Events (SAEs)

An AE is treated as a SAE if the seriousness was classified as "serious".

#### (3) Adverse Drug Reaction

An AE is considered "adverse drug reaction" if the relationship to the investigational product was assessed to be "reasonable possibility".

#### (4) Time to Adverse Events

Time to Adverse Events (days) = AE start date – date of administration in the period of AE occurrence + 1

#### (5) Duration of Adverse Events

Duration of Adverse Events (days) = AE stop date – AE start date + 1

#### (6) Period of Adverse Events occurrence

AEs will be assigned to the last administration of the investigational product before the occurrence.

Period I: AEs occurred on or after the time of administration in Period I but before the time of administration in Period II

Period II: AEs occurred on or after the time of administration in Period II but before the completion of end-of-study assessment.

#### 7.1.2.2 Laboratory Tests

(1) Clinically relevant values flag

Clinically relevant values flag will be attached to the values out of normal range. (L=Lower than normal range, H=Higher than normal range or A=Abnormal).

(2) Laboratory test values below the limit of quantification

Any BLQ data will be treated as LLOQ/2 in summary statistics.

#### 7.1.2.3 12-Lead ECG

(1) Criteria for pre-defined limit

12-lead ECG:

- QTcF > 500 msec
- -500 >= QTcF > 480msec
- -480 >= QTcF > 450msec
- QTcF <= 450 msec
- Change from baseline in QTcF > 60 msec
- Change from baseline in QTcF > 30 msec

#### 7.1.3 Pharmacokinetics Evaluation

#### 7.1.3.1 Plasma Concentration

For the calculation of the summary statistics, concentration values reported as BLQ will be set to 0. In figures, concentration values reported as BLQ will be plotted as 0 in linear scale and not plotted in semi-logarithmic scale.

#### 7.1.3.2 Pharmacokinetic Parameters

For the calculation of PK parameters, actual sampling time (in hours rounded to 3 decimal places) relative to dosing should be used. If the sampling was performed before dosing, time after dosing will be set to 0. When  $k_{el}$  is missing (or cannot be determined),  $t_{1/2}$ ,  $AUC_{0-\infty}$ ,  $AUC_{0-\infty}$ , CL/F, MRT,  $V_z/F$  and  $V_{ss}/F$  will not be calculated.

#### (1) Below the limit of quantification

Concentration below the limit of quantification (BLQ) will be set to 0.

#### (2) Calculation of AUC

Timepoints with missing concentration data will be ignored. Concentration value at the end time of partial AUC will be calculated by linear-linear trapezoidal rule or by extrapolation using elimination rate constant, if there is no valid data exactly at the time.

#### (3) Calculation of V<sub>ss</sub>/F

Pharmacokinetic parameter of V<sub>ss</sub>/F will be calculated as follows:

$$V_{ss}/F = MRT \times CL/F$$

#### 7.2 Analysis Visit Definitions

#### (1) Non-PK related

Analysis visit window is not defined. By-visit summaries will be based on nominal visit or timepoint.

Study day is the relative day to the first treatment. Day -1 is the day before the first treatment, Day 1 is the day of the first treatment, and Day 2 is the next day.

Except for laboratory tests, Day 1 pre dose will be the baseline for Period I and Day 4 pre dose will be the baseline for Period II. For laboratory tests, Day -1 will be the baseline.

#### (2) PK related

Analysis time point and allowable range is defined below.

| Analysis Time Point | Window |
|-----------------------------------------------|-----------------------------|
| Predose | Within 60 min before dosing |
| 0.083 h | Nominal time ± 1 min |
| 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12 h | Nominal time ± 5 min |
| 24, 36, 48 h | Nominal time ± 15 min |

#### 7.3 Data Handling Convention for Missing Data

#### (1) Non-PK related

#### Adverse events:

If severity or relationship should be missing, the most severe or more related category will be imputed for the summary.

#### Other safety:

For safety summaries, only observed data will be used. Unless otherwise specified, missing safety data will not be imputed.

#### (2) PK related

For PK summaries, only observed data will be used. Missing plasma concentration data will not be imputed.

#### 8 STATISTICAL METHODOLOGY

#### 8.1 Study Subjects

#### 8.1.1 Subject Disposition

Subject disposition will be summarized and listed on the randomized subjects.

Randomization details will be listed on the randomized population.

#### 8.1.2 Analysis Populations

Analysis populations will be summarized and listed on the randomized subjects.

#### 8.1.3 Study Drug Exposure

Exposure data will be summarized and listed on the SAF.

#### 8.1.4 Demographic and Other Baseline Characteristics

The following demographic and other baseline characteristics will be used.

| | Categorical | Descriptive |
|-----------------------------|-------------------------------|-------------|
| Sex | Male, Female | |
| Age (years) | | Yes |
| Height (cm) | | Yes |
| Weight (kg) | | Yes |
| BMI (kg/m <sup>2</sup> ) | | Yes |
| Race | Japanese | |
| Medical history | No, Yes | |
| Complication | No, Yes | |
| Concomitant medication* | No, Yes | |
| Allergic history (including | No, Yes | |
| drug allergies) | | |
| Drinking status | No ('Never'), Yes (otherwise) | |
| Smoking status | No ('Never'), Yes (otherwise) | |

<sup>\*</sup> The surface anesthesia for nasogastric tube insertion will be excluded.

Demographic and other baseline characteristics will be summarized and listed on the SAF.

#### 8.1.5 Medical History

Medical history, complication and allergic history will be listed on the SAF.

#### 8.1.6 Concomitant Medications

Concomitant medication will be listed on the SAF.

#### 8.2 Safety Assessments

All safety assessments will be performed on the SAF.

#### 8.2.1 Adverse Events

Overall occurrence of AEs will be summarized using the following categories by treatment.

- Subjects with at least one AE
- Subjects with at least one adverse drug reaction
- Subjects with at least one SAE
- Subjects with at least one serious adverse drug reaction
- Subjects with at least one AE leading to discontinuation of study drug
- Subjects with AE leading to death

The following summaries will also be presented by treatment.

- AEs by SOC and PT
- Adverse drug reactions by SOC and PT
- AEs by SOC, PT and severity

These will be subject-based summaries - multiple occurrences of the event with the same SOC and/or PT within a subject will be counted once in the summaries by SOC and PT; multiple occurrences of the event with the same SOC and/or PT but different severity within a subject will be counted once in the maximum severity category (severe > moderate > mild).

To summarize by treatment, the AE occurred under PO/NGT treatment period will be counted as PO/NGT treatment. Period of AE occurrence is defined in 7.1.2.1 (6).

The followings will be listed.

- AE
- SAE

## 8.2.2 Laboratory Tests

For quantitative tests (i.e. hematology, biochemistry and coagulation), absolute values and changes from baseline will be summarized descriptively by group and visit.

For qualitative tests of urinalysis, number and percentage will be presented by group and visit. Changes from baseline to each visit will be presented as shift-table by group.

All data will be listed.

Below is a list of the laboratory test.

| <b>Laboratory Test</b> | Parameters |
|---|---|
| Hematology | Hemoglobin, hematocrit, RBC count, WBC count, platelet count, MCH, MCHC, MCV, differential white blood count |
| Biochemistry | Na, K, Cl, Ca, inorganic phosphorus, urea nitrogen, creatinine, uric acid, total bilirubin, direct bilirubin, ALT, AST, γ-GTP, ALP, LDH, CK, amylase, total cholesterol, triglycerides, LDL-C, HDL-C, total protein, albumin, glucose, CRP |
| Coagulation test | Prothrombin time, APTT, INR*, prothrombin activity* |
| Urinalysis | Qualitative tests (pH, specific gravity, protein, glucose, occult blood, urobilinogen, bilirubin, ketones), sediment* |

<sup>\*</sup> Only for listing. Not summarized.

#### 8.2.3 Vital Signs

Absolute values and changes from baseline will be summarized for the following parameters by treatment and time point.

- Systolic blood pressure (mmHg)
- Diastolic blood pressure (mmHg)
- Pulse rate (bpm)
- Body temperature (°C)

All data will be listed.

#### **8.2.4** 12-Lead ECGs

Absolute values and changes from baseline will be summarized for the following parameters by treatment and time point.

- Heart rate (bpm)
- PR (msec)
- RR (msec)
- QRS (msec)
- QT (msec)
- QTcF (msec)

For interpretation, number and percentage will be presented by treatment and time point. The percentage of subjects with values outside pre-defined limits will be summarized by treatment and time point.

All data (including interpretation and findings) will be listed.

#### 8.2.5 Physical Examinations

Physical examination will be listed.

#### 8.3 Pharmacokinetics Evaluation

Pharmacokinetic analysis will be performed on the PKPOP. Summaries of concentrations, PK parameters and statistical analysis for unchanged edaravone will be performed using data from subjects whose PK data will be available in both treatments.

#### 8.3.1 Plasma Concentrations and Pharmacokinetic Parameters

(1) Summary tables and listings

Plasma concentrations of unchanged edaravone will be summarized by analysis time point and treatment. All plasma concentrations will also be listed.

(2) Plots of individual plasma concentrations

Individual plasma concentrations vs. actual time for unchanged edaravone will be plotted on both linear/linear and log/linear scales, both by treatment and by subject.

#### (3) Plots of mean plasma concentrations

Mean (+SD) plasma concentrations vs. nominal time curves will be plotted on both linear/linear and log/linear scales superimposing the treatments.

#### 8.3.2 Pharmacokinetic Parameters

The PK parameters listed in Section 2.1.2 will be calculated for each subject using non-compartmental model. Calculations of the parameters, including supplementary parameters, are described in Appendix 1.

The PK parameters will be summarized by treatment and listed. The supplementary parameters will not be summarized but will be included in listing.

#### 8.3.3 Analysis of Variance

AUC<sub>0-t</sub>, AUC<sub>0- $\infty$ </sub> and C<sub>max</sub> of unchanged edaravone will be log transformed and analysed. Only subjects with the parameter value under both treatments will be analysed. Analysis of variance (ANOVA) will be used for analysis. Group, treatment, period and subject (nested in group) will be set to factors. Least squares (LS) means for each treatment will be calculated. These values will be back-transformed and shown in table. The difference of LS means between treatments (nasogastric administration minus oral administration) and 90% CI will be calculated. These values will be back-transformed, so that they show the ratio and 90% CI of PK parameters for nasogastric administration compared to oral administration.

As reference, the other pharmacokinetic parameters of unchanged edaravone will be analysed in the same way, although  $t_{max}$  will not be log transformed prior to the analysis.

# 9 DATA PRESENTATION CONVENTIONS

## 9.1 Number of Digits to Report

#### (1) Non-PK related

| Statistic | Specification | Apply to |
|---|---|---|
| Minimum, Maximum | Same number of DPs as provided in the datasets | All original data (i.e. non-derived) |
| | see section 7.3 | All derived data |
| Mean, SD, Median | One more DP than above | All |
| Percentages <sup>1</sup> | 1 DP | All |

<sup>&</sup>lt;sup>1</sup> Percentages: use 1 place beyond the decimal point, except for the following cases:

#### (2) PK Plasma Concentration

| Statistic | Specification |
|-------------------|---------------------------------------------------|
| Individual value | With the number of DPs to which they are reported |
| Mean, SD, Median, | Same number of DPs as the individual value |
| Minimum, Maximum | |
| CV% | 1 DP |

#### (3) PK Parameters

| Statistic | Specification |
|---|---|
| Individual value | C <sub>max</sub> : same number of DPs as the plasma concentration |
| | AUC%ex: 3DPs |
| | t <sub>max</sub> , lower/upper limit of k <sub>el</sub> : 3 DPs |
| | Adjusted R <sup>2</sup> : 3 DPs |
| | Number of kel points: integer |
| | Other parameters: number of DPs at which minimum |
| · | value of the parameter comes to 3 significant digits. |
| Mean, SD, Median, | Same number of DPs as the individual values |
| Minimum, Maximum, | |
| Geometric mean, LS mean, | |
| Geometric LS mean, CI | |
| CV%, Geometric CV% | 1 DP |
| Ratios | 3 DPs |

If the percentage is equal to 0, then not shown as "(0)" but left blank

If the percentage is equal to 100, then shown as "(100)" without a decimal

# 9.2 Treatments and Groups to Report

| Treatment | For TFLs |
|----------------------------------------------|----------|
| Oral administration of edaravone oral | PO |
| suspension 105 mg | |
| Nasogastric administration of edaravone oral | NGT |
| suspension 105 mg | |

| Group | For TFLs |
|--------------------------------------|----------|
| Oral administration precedent | PO - NGT |
| Nasogastric administration precedent | NGT - PO |

# 9.3 Period, Visit and Time Point to Report

# (1) Non-PK related

Safety:

| D . 16 | ¥7° .*4 € | Time Point Apply to | | | |
|---|---|---|---|---|---|
| Period for<br>TFLs | Visit for<br>TFLs | Time Point<br>for TFLs | Laboratory<br>Tests | Vital Signs | 12-Lead<br>ECGs |
| Screening | Screening | | X | X | X |
| Period 1 | Day -1 | | X | X | X |
| | Day 1 | Pre-dose | | X | X |
| | Day 1 | 1 h | | X | X |
| | Day 2 | 24 h | | X | X |
| | Day 3 | 48 h | X | X | X |
| Period 2 | Day 4 | Pre-dose | | X | X |
| | Day 4 | 1 h | | X | X |
| | Day 5 | 24 h | | X | X |
| | Day 6 | 48 h | X | X | X |
| End of study | End of study | | X | X | X |

Unscheduled tests and tests on discontinuation will not be included in by-visit summaries but will be shown in listings.

# (2) PK-related

| Analysis Visit | Analysis Time Point |
|---|---|
| Day 1 | Pre-dose, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12 h |
| Day 2 | 24, 36 h |
| Day 3 | 48 h |
| Day 4 | Pre-dose, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12 h |
| Day 5 | 24, 36 h |
| Day 6 | 48 h |

#### 10 CHANGE FROM THE PROTOCOL

Geometric CV% will be calculated as a summary statistic for PK parameters instead of 95% CI of geometric mean, and also CV% is added.

90% CI of geometric LS means of PK parameters will not be calculated. The ratio of geometric LS means will be accompanied by 90% CI.

Summary for laboratory tests will be performed not by treatment but by group because there is no baseline for laboratory tests in Period II.

INR and prothrombin activity are added to coagulation test because these results are reported from the laboratory. Whereas hCG is excluded from urinalysis because the results are not collected.

# 11 SOFTWARE

All statistical analyses will be performed using SAS version 9.4 or higher.

The PK parameters will be calculated using WinNonlin® software (version 6.3 or later).

# 12 REFERENCES

N/A

# APPENDIX 1 PHARMACOKINETIC PARAMETER CALCULATIONS

| PK Parameter Calculations | | |
|---|---|---|
| Parameters Unit Calculation | | |
| AUC <sub>0-t</sub> | ng·h/mL | AUC will be calculated using the linear trapezoidal method and actual times |
| | | $AUC_{t_0-t_n} = \sum_{i=1}^{t_n} \frac{t_i - t_{i-1}}{2} (C_{i-1} + C_i)$ |
| | | $AUC_{0-t}$ will be calculated as $AUC$ when $t_0$ is set to time zero and $t_n$ is set to t (the last quantifiable concentration time point). |
| AUC <sub>0-∞</sub> | ng·h/mL | $AUC_{0-\infty} = AUC_{0-t} + C_{last} / k_{el}$<br>$C_{last}$ : last measurable concentration |
| AUC%ex * | % | $AUC\%_{ex} = (AUC_{0-\infty} - AUC_{0-t}) / AUC_{0-\infty} \times 100$ |
| AUC <sub>0-24</sub> | ng·h/mL | will be calculated using time until 24 h drug concentration |
| $C_{max}$ | ng/mL | will be determined by visual inspection |
| t <sub>max</sub> | h | Measured time of C <sub>max</sub> |
| t <sub>1/2</sub> | h | $t_{1/2}$ will be determined as: $t_{1/2} = \log_e(2) / k_{el}$ |
| k <sub>el</sub> | 1/h | The exponential rate constant of the terminal phase, $k_{el}$ , will be estimated by log-linear regression, if determinable. The number of data points included in the regression will be determined by visual inspection. Wherever possible, a minimum of 3 data points will be used in the estimation of $k_{el}$ . During the analysis, this calculation method repeats regressions using the last three points with non-zero concentrations, then the last four points, last five, etc. The time of maximum concentration ( $t_{max}$ ) will be excluded from the estimation of $k_{el}$ . Points with a value of zero for the dependent variable are excluded. For each regression, an adjusted $R^2$ is computed Adjusted $R^2 = 1 - \frac{(1 - R^2) \times (n - 1)}{(n - 2)}$ |
| CL/F<br>MRT | L/h<br>h | where n is the number of data points in the regression and $R^2$ is the square of the correlation coefficient. The regression with the largest adjusted $R^2$ is selected to estimate $k_{el}$ , with these caveats: If the adjusted $R^2$ does not improve, but is within 0.0001 of the largest adjusted $R^2$ value, the regression with the larger number of points is used. $k_{el}$ must be positive, and calculated from at least three data points. $CL/F = Dose / AUC_{0-\infty}$ MRT = $AUMC_{0-\infty} / AUC_{0-\infty}$ AUMC <sub>0-\infty</sub> : area under the first moment curve extrapolated to infinity |

| PK Parameter Calculations | | |
|---|---|---|
| Parameters | Unit | Calculation |
| V₂/F | L | $V_z/F = CL/F \times \frac{1}{k_{el}}$ |
| V <sub>ss</sub> /F | L | $V_{ss}/F = MRT_{po} \times CL/F$ |
| Adjusted R <sup>2</sup> * | T- | Refer to calculation of kel. |
| Number of kel points* | _ | will be determined using number of points used in computing kel. If kel cannot be estimated, zero. |
| Lower limit of kel* | h | will be determined using lower limit on time to be included in the calculation of $k_{\rm el}$ . |
| Upper limit of kel* | h | will be determined using upper limit on time to be included in the calculation of kel. |

<sup>\*</sup> Supplementary parameters.